CLINICAL TRIAL: NCT04925674
Title: Phase Ic Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HEC53856 Capsules in Subjects With Renal Anemia on Dialysis
Brief Title: Study of HEC53856 in Patients With Subjects With End-Stage Renal Disease Receiving Dialysis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Collaborators: Nicoya Therapeutics (Shanghai) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEC53856-RAD-103
Record Dates: First submitted 2021-05-30; First posted 2021-06-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2021-06

CONDITIONS: Hemodialysis; Peritoneal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HEC53856 (Experimental): HEC53856 Oral TIW There will be a total of 3 dose cohorts in the hemodialysis: 100mg，150mg，200mg； There will be only one dose cohort in the peritoneal dialysisp:100mg.
  Interventions: Drug: HEC53856

INTERVENTIONS:
Drug: HEC53856 — The 100mg dose cohort in the hemodialysis: D1 single oral administration of the investigation product 2.5h before hemodialysis; Three times a week for 6 weeks starting from D8, oral administration of the test drug 2.5h after hemodialysis.
  The rest dose cohorts in the hemodialysis: Three times a week for 6 weeks starting from D1, oral administration of the investigation product 2.5h after hemodialysis.
  The dose cohort in the peritoneal dialysis: Three times a week for 6 weeks starting from D1, oral administration of the investigation product after fasting.

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of HEC53856 capsules on anemia in subjects with chronic kidney disease on dialysis.

DETAILED DESCRIPTION:
The purpose of this multicenter, open-label, dose-increasing, multiple-dose study was to evaluate the safety, tolerability,PK and preliminary efficacy of HEC53856 capsules in renal anemia subjects on dialysis.

The study consists of two parts, hemodialysis or peritoneal dialysis . Within each part participants will be administrated for HEC53856.

There are three study periods:

Screening period :up to 2weeks; Treatment period: 6 weeks（except that 7 weeks in the 100mg cohort in the hemodialysis）; Follow-up period: 2weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily participated in this clinical trial and signed an informed consent form;
2. 18-70 years old, weight 45~90kg, including cut-off value;
3. Hemodialysis (Hemodialysis, HD): Patients with end-stage renal disease who are on stable dialysis receive 3 times a week hemodialysis for at least 3 months before screening, and can receive 3 times a week hemodialysis at regular intervals during the test. The duration of the subject's hemodialysis treatment must be 3-4.5 hours (including the cut-off value); Peritoneal dialysis: For patients with end-stage renal disease on stable dialysis, the subject must receive peritoneal dialysis for at least 3 months before screening;
4. Subjects stop EPO 14 days or 5 half-lives (whichever is the longest) before taking the test drug for the first time;
5. Subjects have stable dialysis methods and dialysis prescriptions, and are expected to have no major treatment changes or no drastic changes in their condition during the clinical trial period;
6. During the screening period, the hemoglobin value obtained by the two tests of Visit 1 and Visit 2 must be > or = 8.0 g/dL and <11.0 g/dL, and the difference between the two must be < or = 1.5 g/dL.

Exclusion Criteria:

1. Existence of past medical history or conditions that may cause anemia other than nephropathy, including but not limited to blood system diseases, such as thalassemia, aplastic anemia, hemolytic anemia, multiple myeloma, myelodysplastic syndrome, etc.; Autoimmune diseases that may affect red blood cell production, such as systemic lupus erythematosus, rheumatoid arthritis, etc.; Bleeding diseases, such as gastrointestinal bleeding, obstetrics and gynecology bleeding diseases, etc.
2. During the study period, those who plan to change the dialysis method/mode or the flux of the hemodialysis machine, such as changing from peritoneal dialysis to hemodialysis
3. Those who have any of the following heart/cerebrovascular diseases:

   1. Acute coronary syndrome, stroke (except lacunar infarction) or thromboembolic disease (such as deep vein thrombosis or pulmonary embolism) occurred within 6 months before screening;
   2. Heart Function III of New York Society of Cardiology Or grade IV congestive heart failure, or severe arrhythmia, including but not limited to ventricular tachycardia, ventricular fibrillation, III degree atrioventricular block, etc.
4. Those who have any of the following medical or surgical history:

   1. Those who plan to undergo major surgery 3 months before screening or during the study period (except for hemodialysis access repair) or blood transfusion therapy;
   2. Have peritoneal dialysis related 3 months before screening Peritonitis, history of infection or leakage of peritoneal tube tunnel;
   3. history of malignant tumor within 5 years prior to screening (except for cured skin basal cell carcinoma and cervical carcinoma in situ), or current assessment of potential malignant tumor;
   4. suffering Uncontrollable or symptomatic secondary hyperparathyroidism, plasma iPTH>800pg/ml;
   5. History of dysphagia or any gastrointestinal disease that affects drug absorption, history of gastric/jejunum/colon resection; f ) Those who have a serious infection and are receiving systemic antibiotic treatment;

   g) Anyone who has participated or plans to participate in an organ transplant within 6 months; h) Have a history of chronic liver disease (such as: chronic infectious hepatitis, chronic autoimmune liver disease, cirrhosis Or liver fibrosis); i) Patients with a history of polycystic kidney disease.
5. Any of the following laboratory abnormalities during the screening period:

   1. Folic acid <6.8nmol/L (3ng/ml) and/or VitB12<74pmol/L (100ng/ml);
   2. Serum albumin <3 g/dL;
   3. AIDS antibody , Treponema pallidum antibody, hepatitis B surface antigen or hepatitis C antibody positive for any one;
   4. ALT>3×ULN and/or AST>3×ULN, or total bilirubin>1.5× ULN;
6. Subjects received intravenous iron supplementation within 4 weeks before screening, or used Chinese patent medicines, androgens and anabolic hormone drugs, hypoxia-inducible factor prolyl hydroxylase for the treatment of anemia within 4 weeks before screening Inhibitors (such as Roxastat capsules) and other drugs (except ESAs and their derivatives, oral irons, stable oral irons can be taken within 4 weeks before the screening, and in the screening period and after the start of the trial drug Continue to take the fixed dose for 6 weeks.)
7. Subjects who are expected to take BCRP inhibitors, BCRP inducers, CYP2C8 inhibitors and inducers within 14 days before taking the test drug (or 5 half-lives of the drug, whichever is the longest) until the end of the drug;
8. Those who have a history of drug abuse or drug abuse within 6 months before screening;
9. The mean systolic blood pressure =180 mmHg and/or the diastolic blood pressure > or = 110 mmHg of two supine blood pressure measurements at least 1 hour apart during the screening period;
10. People with a history of severe allergic disease or drug allergy, or those who are allergic to test drugs or their excipients;
11. Those who drink more than 14 units per week in the 3 months before screening (1 unit of alcohol ˜ 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine), or those who cannot abstain from alcohol during the hospitalization;
12. Those who smoked more than 10 cigarettes per day in the 3 months before screening, or who could not stop using any tobacco products during the hospitalization;
13. Women who have a positive pregnancy test or are breastfeeding, or men and women who refuse to take effective contraceptive measures within 4 weeks from the signing of the informed consent form to the end of the last trial drug administration;
14. Participated in other clinical trials within 3 months before screening (Definition of participation: accepted experimental drugs or instrument);
15. Subjects may not be able to complete all research visits or procedures required by the research protocol, and/or fail to comply with all required research procedures;
16. The investigator believes that there are other factors that are not suitable for participating in this trial;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 2 weeks after last dose
  To assess the safety and tolerability of therapy by incidence of treatment-emergent adverse events after multiple doses of HEC53856 capsule

SECONDARY OUTCOMES:
AUC0-t | Up to 72 hours after single and multiple drug dosing
  Area under the concentration versus time curve (AUC) from time zero to the time of the last quantifiable concentration
Cmax | Up to 72 hours after single and multiple drug dosing
  Maximum observed plasma concentration
Tmax | Up to 72 hours after single and multiple drug dosing
  Time of the maximum observed plasma concentration
T½ | Up to 72 hours after single and multiple drug dosing
  Apparent terminal elimination half-life
Vz/F | Up to 72 hours after single and multiple drug dosing
  Apparent volume of distribution
Changes in mean hemoglobin | Up to 2 weeks after the last dose
  Changes in mean hemoglobin (Hb) relative to baseline during visit 8 and 9.
Hemoglobin response | Up to 2 weeks after the last dose
  Percentage of subjects who met the hemoglobin response after dosing
E-AUC0-t | Up to 72 hours after single and multiple drug dosing
  Area under the EPO concentration versus time curve (AUC) from time zero to the time of the last quantifiable concentration
Emax | Up to 72 hours after single and multiple drug dosing
  Maximum observed EPO concentration
E-Tmax | Up to 72 hours after single and multiple drug dosing
  Time of the maximum observed EPO concentration
Serum lipid | week 6
  Changes in Serum lipid relative to baseline at visit 8.
Indicators of iron | week 6
  Changes in the Indicators of iron relative to baseline at visit 8
High-sensitivity C-reactive protein | week 6
  Changes in the High-sensitivity C-reactive protein relative to baseline at visit 8.
Reticulocytes | Up to week 8
  Changes in the mean Reticulocytes relative to baseline after doses.
VEGF | week 6
  Changes in the VEGF relative to baseline after doses.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sichuan Provincial People's Hospital, Chengdu
  - The First Affiliated Hospital of Shantou University Medical College, Shantou
  - The First Hospital of China Medical University, Shenyang
  - General Hospital of Tianjin Medical University, Tianjin
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang
  - The Fifth Affiliated Hospital Sun Yat-sen University, Zhuhai